CLINICAL TRIAL: NCT05399030
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Single and Multiple Ascending Dose Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ICP-332 in Healthy Subjects
Brief Title: A Phase I Randomized, Double-Blind, Placebo-Controlled, Parallel Group Clinical Study of ICP-332 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: ICP-CL-00601
Record Dates: First submitted 2022-05-22; First posted 2022-06-01 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICP-332 (Experimental): Single ascending doses of ICP-332 tablet; Multiple ascending doses of ICP-332 tablet
  Interventions: Drug: ICP-332
- Placebo (Placebo Comparator): Single ascending doses of placebo; Multiple ascending doses of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ICP-332 — ICP-332 will be administered as tablet
  Arms: ICP-332
Other: Placebo — Matching placebo will be administered as tablet
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel group, single and multiple ascending dose phase I study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of ICP-332 in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) between 18-26 kg/m2, the weight of male subject should not be less than 50 kg, and the weight of female subject should not be less than 45 kg.
2. Age and fertility status

   1. Male or infertile female subjects who are between 18-45 years old (inclusive).
   2. Female subjects who are infertile.
   3. Male subjects and their partners must agree to use effective contraception.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic and other diseases, or allergic diseases.
2. Subjects with clinically significant gastrointestinal dysfunction that may affect drug intake, transport or absorption.
3. Acute disease state (such as nausea, vomiting, pyrexia or diarrhea, etc.) within 14 days before administration.
4. Other situations judged by the investigator to be unsuitable to join this trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-08-14 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment-Emergent Adverse Events (AEs). | Baseline up to 28 days after last dose.

SECONDARY OUTCOMES:
Change from baseline in Maximum concentration (Cmax) | Single ascending dose: baseline up to 72 hours; post-dose multiple ascending dose: baseline to Day 14.
Change from baseline in blood cells. | Multiple ascending dose: Baseline to 28 days.
  measuraments (e.g. blood biochemistry tests, hematology, coagulation tests); outcome measure (e.g. absolute blood cells count)

CONTACTS AND LOCATIONS:
Overall Officials: Qing Wen, Principal Investigator — Jinan Central Hospital
Locations (1):
- Jinan Central Hospital, Jinan, China